CLINICAL TRIAL: NCT06531811
Title: A Randomized, Open-label, Single-dose, 2-Treatment, 2-Period, Crossover Study to Assess the Relative Bioavailability of AZD8630 Following a Device and Formulation Transition in Healthy Participants.
Brief Title: A Study to Investigate the Relative Bioavailability of AZD8630 Following a Device and Formulation Transition in Healthy Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: D6830C00002
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Healthy Participants
Keywords: Trehalose/leucine/trileucine/citrate (TLTC); Trehalose/leucine/trileucine/histidine (TLTH); Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: This is an open-label, 2-period cross over study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Sequence 1 (Treatment A- Treatment B) (Experimental): Participants will receive Treatment A (AZD8630 Monodose inhalation powder) crossover to Treatment B (AZD8630 test inhalation powder)
  Interventions: Drug: AZD8630 (test formulation) via test inhaler; Drug: AZD8630 (reference formulation) via Monodose inhaler; Device: Test inhaler; Device: Monodose inhaler
- Sequence 2 (Treatment B- Treatment A) (Experimental): Participants will receive Treatment B (AZD8630 test inhalation powder) crossover to Treatment A (AZD8630 Monodose inhalation powder)
  Interventions: Drug: AZD8630 (test formulation) via test inhaler; Drug: AZD8630 (reference formulation) via Monodose inhaler; Device: Test inhaler; Device: Monodose inhaler

INTERVENTIONS:
Drug: AZD8630 (test formulation) via test inhaler — Participants will receive AZD8630 via test inhaler.
Drug: AZD8630 (reference formulation) via Monodose inhaler — Participants will receive AZD8630 via Monodose inhaler.
Device: Test inhaler — Participants will receive AZD8630 via test inhaler.
Device: Monodose inhaler — Participants will receive AZD8630 via Monodose inhaler.

SUMMARY:
The purpose of this study is to evaluate the potential difference between pharmacokinetics (PK), safety, tolerability and device performance between the AZD8630 test formulation and the AZD8630 reference formulation.

DETAILED DESCRIPTION:
This is a randomized, open-label, 2- treatment, 2- period study with a duration of approximately 6 weeks.

The Study will comprise of:

* A Screening period of 28 days,
* Treatment Period 1 on Day 1 and Treatment Period 2 on Day 9
* A Follow-up visit within 7 days (± 2 days) after the last dose in Period 2.

Participants will be randomized 1:1 to either Sequence 1 or Sequence 2.

* Sequence 1: Treatment A (AZD8630 Monodose inhalation powder) crossover to Treatment B (AZD8630 test inhalation powder).
* Sequence 2: Treatment B (AZD8630 test inhalation powder) crossover to Treatment A (AZD8630 Monodose inhalation powder).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Healthy participants aged 18-55 years with suitable veins for cannulation or repeated venipuncture.
* Females participants of childbearing potential must not be lactating and, if sexually active, agree to use highly effective contraception from time of first administration of study intervention until 20 days after last dose of study intervention.
* All females must have a negative serum pregnancy test and must at the Screening Visit.
* Sexually active male participants and their partners of childbearing potential must be willing to use highly effective contraception measures from the time of first administration of study intervention administration until 20 days after the last dose of study intervention and on admission
* Healthy participants must have a FEV1 ≥ 80% of the predicted value regarding age, height, gender, and ethnicity at the Screening Visit.
* Have a BMI between 18 and 32 kg/m2 inclusive and weigh at least 45 kg.

Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study intervention.
* History of any upper or lower respiratory tract infection in the 14 days before screening or during the Screening Period.
* Clinically significant history of atopy or allergy to common allergens including house dust mite and pollens, or a history of childhood asthma, as judged by the investigator.
* Medical history of or treatment for hepatitis B or hepatitis C.
* Other latent or chronic infections (e.g., recurrent sinusitis, genital or ocular herpes, or urinary tract infections) or at risk of infection (major surgery, major trauma, or significant infection) within 90 days of screening, or history of skin abscesses withing 90 days of screening.
* History of cancer within the last 10 years (20 years for breast cancer) except for basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix treated and considered cured. Any history of lymphoma is not allowed.
* Have received live, live attenuated or messenger ribonucleic acid vaccine in the 4 weeks prior to Screening Visit.
* History of or ongoing acquired or inherited immunodeficiency disorders including but not limited to HIV, common variable immunodeficiency or taking immune replacement therapy.
* A helminth parasitic infection diagnosed within 24 weeks of Visit 1 that has not been treated or has not responded to standard of care therapy.
* Any laboratory values with the following deviations at the Screening Visit or on admission to the Clinical Unit.
* Any clinically important abnormalities in clinical chemistry or hematology results at screening and/or admission to the Clinical Unit, as judged by the investigator.
* Abnormal vital signs, after 5 minutes supine rest, at screening and/or admission to the Clinical Unit.
* Any clinically important abnormalities in rhythm, conduction, or morphology of the resting 12-lead ECG, at screening and/or admission to the Clinical Unit, as judged by the investigator that may interfere with the interpretation of QTc interval changes, a prolonged PR interval and abnormal ST wave morphology.
* Current smokers or those who have smoked or used nicotine products or inhalational cannabis/marijuana products (including e-cigarettes) within the previous 6 months prior to screening or has smoking history of > 10 pack years. Known or suspected history of alcohol.
* Known or suspected history of alcohol or drug abuse (including cannabis/marijuana products) or excessive intake of alcohol as judged by the investigator. The use of oral cannabis is permitted.
* Positive screen for drugs of abuse (including any cannabis/marijuana products), or alcohol or cotinine (nicotine) at screening or on admission to the Clinical Unit.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the investigator.
* History of hypersensitivity or anaphylaxis to any components of AZD8630 formulation.
* History of documented immune complex disease (Type III hypersensitivity reactions) to mAb administration.
* Receipt of immunoglobulin or blood products within 4 weeks prior to Screening Visit.
* Excessive intake of caffeine-containing drinks or food (eg, coffee, tea, chocolate) defined as the regular consumption of more than 500 mg of caffeine per day (eg, > 5 cups of coffee [one cup ~100 mg caffeine]; one cup of tea ~30 mg caffeine) or would likely be unable to refrain from the use of caffeine-containing beverages during confinement at the investigational site.
* Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the first administration of study intervention.
* Plasma donation within one month of the Screening Visit or any blood donation/blood loss > 500 mL during the 3 months prior to the Screening Visit.
* Participants who have previously received AZD8630.
* Participants who have medical dietary restrictions or dietary restrictions for which the site are unable to cater.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 30 days of the first administration of study intervention in this study or within 5 half-lives of the medication, whichever is the longest.
* Pregnancy or intention to become pregnant during the study, breastfeeding, or unwillingness to use a highly effective method of contraception throughout the study in female participants of childbearing potential or lactating woman.
* Judgment by the investigator that the participant should not participate in the study if they have any ongoing or recent (i.e., during the Screening Period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
* Vulnerable participants, e.g., kept in detention, protected adults under guardianship

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-08-06 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
Area under the serum concentration-time curve from time zero to the last quantifiable concentration test/Monodose | From Baseline Day 1 to Day 11
  To evaluate the relative bioavailability of AZD8630 test device compared to AZD8630 Monodose device.

SECONDARY OUTCOMES:
Maximum observed plama (peak) drug concentration (Cmax) | From Baseline Day 1 to Day 11
  To evaluate the Cmax of AZD8630 following inhaled administration of the AZD8630 test formulation and the AZD8630 Monodose formulation.
Area under the plasma concentration curve from zero to infinity (AUCinf) | From Baseline Day 1 to Day 11
  To evaluate the AUCinf of AZD8630 following inhaled administration of the AZD8630 test formulation and the AZD8630 Monodose formulation.
Area under the plasma concentration curve from zero to last quantifiable concentration (AUClast) | From Baseline Day 1 to Day 11
  To evaluate the AUClast of AZD8630 following inhaled administration of the AZD8630 test formulation and the AZD8630 Monodose formulation.
Time to reach peak or maximum observed concentration or response following drug administration (tmax) | From Baseline Day 1 to Day 11
  To evaluate the tmax of AZD8630 following inhaled administration of the AZD8630 test formulation and the AZD8630 Monodose formulation.
The last time point at which the concentration is measured (tlast) | From Baseline Day 1 to Day 11
  To evaluate the tlast of AZD8630 following inhaled administration of the AZD8630 test formulation and the AZD8630 Monodose formulation.
Typical elimination rate constant (λz) | From Baseline Day 1 to Day 11
  To evaluate the λz of AZD8630 following inhaled administration of the AZD8630 test formulation and the AZD8630 Monodose formulation.
Half-life associated with terminal slope of a semi-logarithmic concentration time curve (t½λz) | From Baseline Day 1 to Day 11
  To evaluate the t½λz of AZD8630 following inhaled administration of the AZD8630 test formulation and the AZD8630 Monodose formulation.
Area under the plasma concentration curve from zero to 24 (AUC [0-24]) | From Baseline Day 1 to Day 11
  To evaluate the AUC (0-24) of AZD8630 following inhaled administration of the AZD8630 test formulation and the AZD8630 Monodose formulation.
Area under the plasma concentrationcurve from zero to 24, divided by dose (AUC [0-24]/D) | From Baseline Day 1 to Day 11
  To evaluate the (AUC [0-24]/D) of AZD8630 following inhaled administration of the AZD8630 test formulation and the AZD8630 Monodose formulation.
Area under the plasma concentration curve from zero to infinity, divided by dose (AUCinf/D) | From Baseline Day 1 to Day 11
  To evaluate the AUCinf/D of AZD8630 following inhaled administration of the AZD8630 test formulation and the AZD8630 Monodose formulation.
Extrapolated area under the curve from tlast to infinity, expressed as percentage of AUCinf (%AUCextr) | From Baseline Day 1 to Day 11
  To evaluate the %AUCextr of AZD8630 following inhaled administration of the AZD8630 test formulation and the AZD8630 Monodose formulation.
Maximum observed plama (peak) drugconcentration, by dose (Cmax/D) | From Baseline Day 1 to Day 11
  To evaluate the Cmax/D of AZD8630 following inhaled administration of the AZD8630 test formulation and the AZD8630 Monodose formulation.
Apparent total body clearence of drugfrom plasma after extravascularadministration (CL/F) | From Baseline Day 1 to Day 11
  To evaluate the CL/F of AZD8630 following inhaled administration of the AZD8630 test formulation and the AZD8630 Monodose formulation.
Volume of distribution (apparent) at steady state following extravascularadministration based on terminalphase (Vz/F) | From Baseline Day 1 to Day 11
  To evaluate the Vz/F of AZD8630 following inhaled administration of the AZD8630 test formulation and the AZD8630 Monodose formulation.
Number of participants with adverse event (AEs) | From Screening (Day -28) to Follow-up visit (7 days post last dose of AZD8630)
  To further assess the safety and tolerability following single inhaled administration of AZD8630 test formulation and AZD8630 Monodose formulation in healthy participants.
Number of AEs and SAEs associated with test device | From Baseline Day 1 to Day 11
  To assess the safety and performance of the test device.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure."Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/